CLINICAL TRIAL: NCT01006941
Title: Trichuris Suis Ova Therapy for Relapsing Multiple Sclerosis - a Safety Study
Acronym: TRIMS A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Copenhagen (Other); Statens Serum Institut (Other); Copenhagen University Hospital, Hvidovre (Other); OvaMed GmbH (Industry)
Responsible Party: Principal Investigator, Ana Voldsgaard, MD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rigshospitalet, DMSC
Record Dates: First submitted 2009-10-07; First posted 2009-11-03 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Multiple sclerosis; safety; MRI; immunological; Helminths; Trichuris suis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trichuris suis ova (Experimental)
  Interventions: Biological: Trichuris suis ova

INTERVENTIONS:
Biological: Trichuris suis ova — 2500 ova per dose, orally, every second week, during 12 weeks
  Other Names: TSO

SUMMARY:
The hypothesis of this study is that treatment with Trichuris suis ova will be safe and effective as an oral treatment of patients with relapsing multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 55 years
* relapsing course of multiple sclerosis (relapsing-remitting or secondary progressive MS with relapses
* duration of the disease of at least 1 year
* no disease modifying therapy or unchanged immunomodulatory therapy for the last 3 months
* at least 2 documented relapses during the last 24 months with the last relapse within the last 12 months

Exclusion Criteria:

* pregnancy or period of breastfeeding or missing adequate contraceptive protection for female premenopausal patients
* relapse in the last month prior enrolment
* treatment with steroids in the last 30 days
* previous treatment with mitoxantroneduring the last year
* previous treatment with cyclophosphamide or other intensive immunosuppression, total irradiation
* treatment with glatiramer acetate, azathioprine, IVIG or any other immunosuppressive or immunomodulatory drug apart from interferon-beta in the 6 months prior to enrolment
* cardiac insufficiency (NYHA III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, instable or advanced ischemic heart disease (CCS III or IV), malignant hypertension
* diabetes mellitus and other autoimmune diseases
* history of renal insufficiency
* stay in tropical areas during the last 3 months
* eosinophilia in the blood (> 0,45 billion/l)
* concurrent systemic infections

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
MRI activity judged by the number of new or enlarging T2 lesions, number of Gd enhancing lesions and volume of T2 lesions | every 3. week. 3 MRI before treatment and 4 MRI during and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Per S Sørensen, Professor, Study Director — Rigshospitalet, Danish Multiple Slerosis Research Center
Locations (1):
- Danish Multiple Sclerosis Center, Rigshospitalet, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Voldsgaard A, Bager P, Garde E, Akeson P, Leffers AM, Madsen CG, Kapel C, Roepstorff A, Thamsborg SM, Melbye M, Siebner H, Sondergaard HB, Sellebjerg F, Sorensen PS. Trichuris suis ova therapy in relapsing multiple sclerosis is safe but without signals of beneficial effect. Mult Scler. 2015 Nov;21(13):1723-9. doi: 10.1177/1352458514568173. Epub 2015 Feb 19. PMID 25698173